CLINICAL TRIAL: NCT02290626
Title: Randomized Comparison of Elemental Diets and Semi-solid Diets on Gastric Excretion and Gastroesophageal Regurgitation in Bedridden Gastrostomy-fed Patients
Brief Title: Elemental Diets vs. Semi-solid Diets on Gastric Excretion and Gastroesophageal Regurgitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study protocol was changed.
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ED vs. Semi-solid
Record Dates: First submitted 2014-11-02; First posted 2014-11-14 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Gastro-oesophageal Reflux
Keywords: Elemental diet; semi-solid diet; gastric emptying; GER; PEG
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elemental diet (Experimental): Study 1: Elemental diet (300 kcal/300 ml) containing a contrast medium (5 ml) is administered within 15 min using the PEG.
  Study 2: Elemental diet (200 kcal/200 mL) labeled with 100 mg [13C]sodium acetate is administered within 15 min using the PEG.
  Interventions: Drug: Elmental diet
- Semi-solid diet (Active Comparator): Study 1: Semi-solid diet (300 kcal/300 ml) containing a contrast medium (5 ml) is administered within 15 min using the PEG.
  Study 2: Semi-solid diet (200 kcal/200 mL) labeled with 100 mg [13C]sodium acetate is administered within 15 min using the PEG.
  Interventions: Drug: Semi-solid diet

INTERVENTIONS:
Drug: Elmental diet — elemental diet is administered using PEG.
  Other Names: Elental
  Arms: Elemental diet
Drug: Semi-solid diet — Semi-solid diet is administered using PEG.
  Other Names: Racol-NF semisolid
  Arms: Semi-solid diet

SUMMARY:
Study 1: A randomized, crossover trial using elemental or semi-solid diets containing contrast medium as a tracer given to bedridden PEG patients. The distribution of the administered diets is assessed at the distal esophagus, proximal and distal stomach using a plain CT before and 1 hour after the administration.

Study 2: A randomized, crossover trial using elemental or semi-solid diets containing 13C sodium acetate as a tracer given to bedridden PEG patients. 13C breath tests are performed to estimate gastric emptying.

DETAILED DESCRIPTION:
Study 1: A mix of elemental or semi-solid diet (300 kcal/300 mL ) and contrast medium (5ml) is administered using PEG, respectively. Using a plain CT, the distribution of the administered diet is assessed at the distal esophagus, proximal and distal stomach before and 1 hour after the administration. The volume of the residual diet at the distal esophagus, proximal and distal stomach is compared between an elemental and semi-solid diet.

Study 2: Either the elemental diet or semi-solid diet (200 kcal/200 mL) is labeled with 100 mg [13C]sodium acetate (Cambridge Isotope Laboratories Inc, Cambridge, MA) and is administered in the first 15 min of the examination at the same speed using the PEG.

ELIGIBILITY:
Inclusion Criteria:

* Bedridden PEG patients are admitted for fever which is the most common reason for admission of PEG patients to our hospital.

Exclusion Criteria:

* Regular use of gastric acid blockers, motility drugs, benzodiazepines or opioids, any clinical evidence of acute infection, a history of abdominal surgery, and an American Society of Anesthesiologists physical status of class IV or V.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal regurgitation | A half year
  The distribution of the administered diets is assessed at the distal esophagus, proximal and distal stomach using a plain CT before and 1 hour after the administration.

SECONDARY OUTCOMES:
Gastric excretion | A half year
  13C breath tests were performed to estimate gastric excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Japan